CLINICAL TRIAL: NCT06139094
Title: Magnetocardiography as a Noninvasive Diagnostic Strategy for Suspected Myocardial Ischemia With the Absence of Obstructive Coronary Artery Disease As Confirmed by Thermodilution-Derived CFR
Brief Title: MCG for Suspected INOCA Confirmed by Thermodilution-Derived CFR
Acronym: MICRO(T)
Status: Completed | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MICRO(T)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Heart Disease; Coronary Microvascular Disease; Angina
Keywords: Magnetocardiography; CFR via Thermodilution; CardioFlux
MeSH Terms: conditions — Myocardial Ischemia; Microvascular Angina; Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- CMD negative: Participants in this group exhibit no signs of Coronary Microvascular Disease (CMD), as evidenced by a CFR measurement equal to or greater than 2.5. This group serves as the comparative reference, representing individuals without CMD-related myocardial ischemia.
  Interventions: Device: CardioFlux Magnetocardiography
- CMD positive: This group comprises participants demonstrating signs of Coronary Microvascular Disease (CMD), defined by a coronary flow reserve (CFR) measurement of less than 2.5. Participants in this category are experiencing myocardial ischemia without significant blockages in their coronary arteries.
  Interventions: Device: CardioFlux Magnetocardiography

INTERVENTIONS:
Device: CardioFlux Magnetocardiography — The device is a magnetocardiography (MCG) scanner named CardioFlux, which is paired with a cloud processing software. CardioFlux devices are owned by Genetesis and are currently cleared for the acquisition, display, and analysis of magnetic fields generated by cardiac electrical activity (K182571, FDA clearance letter available for download online)

SUMMARY:
This study will be an observational registry to investigate the ability of magnetocardiography (MCG) in determining the presence of myocardial ischemia with the absence of obstructive coronary artery disease, by using an invasive reference standard coronary flow reserve (CFR) measured using thermodilution for diagnosis. The device is a magnetocardiography (MCG) scanner named CardioFlux, which is paired with cloud processing software. A CardioFlux scan appointment shall last approximately 15 minutes in duration and include a patient questionnaire following the scan.

DETAILED DESCRIPTION:
This observational registry study focuses on investigating the efficacy of magnetocardiography (MCG) in detecting myocardial ischemia secondary to coronary microvascular dysfunction (CMD) in the absence of obstructive coronary artery disease. The reference standard for diagnosis will be invasive coronary flow reserve (CFR) measured using thermodilution.

The study utilizes a magnetocardiography (MCG) scanner known as CardioFlux, complemented by cloud processing software. The scanning procedure is designed to last approximately 15 minutes per participant, encompassing 5 minutes for patient preparation, 5 minutes for the CardioFlux scan, and an additional 5 minutes for a post-scan patient survey.

The primary objective is to assess the ability of MCG, through CardioFlux, to accurately determine the presence of myocardial ischemia in comparison to the reference standard CFR. The study will provide valuable insights into the diagnostic potential of MCG and its role in CMD detection, contributing to advancements in non-invasive cardiovascular diagnostics.

The primary study outcome measures shall be the detection of myocardial ischemia with no obstructive coronary artery disease (INOCA) using MCG-CF compared to Cardiac Thermodilution derived CFR. The secondary study outcome measures shall be the MCG Questionnaire, Demographic data (age, sex, height, weight, etc.), Relevant patient medical history, EKG results (if available), and Invasive CFR/angiogram results.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of enrollment.
* Signs and symptoms of coronary ischemia that prompted further evaluation by either invasive coronary angiography or coronary CT angiogram) within the previous 5 years.
* Willing to provide written informed consent.
* Non-obstructive CAD defined as: 0 to 49% diameter reduction of a major epicardial vessel or FFR>0.80 (or non-hyperemic equivalent of iFR or RFR >0.89)
* Completed invasive CFR via thermodilution method within 6 months of informed consent.
* Successfully passing CardioFlux's MCG ""Quality Preview" prior to MCG study scan.

Exclusion Criteria:

* Patients unable to fit into the CardioFlux device.
* Patients who meet device contraindications (as specified in section 1.4 of the protocol) NOTE: Sternotomy wires and stents are typically acceptable.
* Patients unable to lie supine for 5 minutes.
* History of non-ischemic dilated or hypertrophic cardiomyopathy.
* Documented acute coronary syndrome (ACS) within the previous 30 days.
* Known left ventricular ejection fraction (LVEF) <45%, or hospitalization for Reduced ejection fraction within 180 days. (HFpEF is permitted).
* Currently in atrial fibrillation or atrial flutter at the time of enrollment.
* Estimated glomerular filtration rate (eGFR) <30 ml/min.
* Moderate or severe valvular disease (including aortic stenosis or insufficiency).
* Life expectancy <1-yrs. due to non-cardiovascular comorbidity.
* Concurrent enrollment in a clinical trial in which therapeutic intervention is administered within 30 days of enrollment.
* Pregnancy.
* Dextrocardia.
* History of Left or Right Bundle Branch Block within 6 months of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with suspected or confirmed myocardial ischemia with no obstructive coronary artery disease (INOCA).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Detection of Myocardial Ischemia in the Absence of Obstructive Coronary Artery Disease (INOCA) | 6 months
  This observational registry study focuses on investigating the efficacy of magnetocardiography (MCG) in detecting myocardial ischemia secondary to coronary microvascular dysfunction (CMD) in the absence of obstructive coronary artery disease.

SECONDARY OUTCOMES:
Patient-Reported Experiences with MCG | 6 months
Participant Demographic Characteristics | 6 months
  weight (kg)
Participant Demographic Characteristics | 6 months
  age, sex, vital signs
Electrocardiogram (EKG) | 6 months
  If participants have undergone electrocardiogram (EKG) testing, the results will be considered to provide additional insights into their cardiac electrical activity.
Invasive Coronary Flow Reserve (CFR) and Angiogram Outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Odayme E Quesada, MD, Principal Investigator — The Christ Hospital
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Ascension St. John Hospital, Detroit, Michigan
  - The Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No